CLINICAL TRIAL: NCT04824365
Title: Two Week Sub-chronic Double-blinded Placebo Controlled Trial Designed to Determine if Sodium Pyruvate Nasal Spray Will Reduce the Symptoms, Duration and Replication of COVID-19 Infection
Brief Title: Sodium Pyruvate Nasal Spray Treatment of COVID-19 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cellular Sciences, inc. (Industry)
Collaborators: Missouri State University (Other); Dynamic DNA Laboratories (Industry); Trinity Health System (Industry); Family First Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSI-COVID-19_007
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Results first posted 2022-09-26 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BASS2 protein, Arabidopsis; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 15 COVID-19 infected patients will be assigned to the placebo and 15 COVID-19 infected patients assigned to the drug treatment for a total of 30 patients.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment of COVID-19 infected patients with a sodium pyruvate nasal spray (Experimental): In this arm, patients will be provided with N115 sodium pyruvate nasal spray and instructed to use it 3x daily for 14 days. This group will be compared to the placebo control group to determine if sodium pyruvate reduces the symptoms, duration and replication of COVID-19 infection.
  Interventions: Drug: Sodium Pyruvate
- Placebo control treatment of COVID-19 infected patients (Placebo Comparator): In this arm, patients will be provided with a saline nasal spray as a placebo control. Patients will use the saline nasal spray 3x daily for 14 days, similar to the sodium pyruvate drug arm. This will serve as a control for the symptoms, duration and replication of COVID-19 infection.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Sodium Pyruvate — Subjects will use a sodium pyruvate nasal spray 3x daily for 14 days.
  Other Names: N115
  Arms: Treatment of COVID-19 infected patients with a sodium pyruvate nasal spray
Other: Saline — Subjects will use a saline nasal spray 3x daily for 14 days.
  Arms: Placebo control treatment of COVID-19 infected patients

SUMMARY:
Cellular Sciences Inc has submitted over 17 human clinicals (phase I, II, III including animal safety data) to the FDA for the reduction of respiratory inflammation and inflammatory cytokines including IL-6 the cause of the cytokine storm in COVID patients. These clinicals demonstrated a reduction of inflammation in all lung and sinus diseases, in patients with COPD, Pulmonary fibrosis, CF, asthma, sinusitis , the flu and nasal inflammation and congestion. Inhaled sodium pyruvate reduces inflammation, congestion and in our phase III clinical study with Idiopathic Pulmonary Fibrosis patients we demonstrated statistically and clinical significant increase in FEV-1, SaO2, FVC, FEV-1/FVC ratios (form 52% to 86%) and a decrease in hypoxemia, and a reduction in coughing. Inhaled sodium pyruvate alleviated the symptoms associated with COVID-19 patients in Pulmonary Fibrosis, and may be a solution to the lingering COVID-19 symptoms in patients that had the COVID-19 infection for example long haulers. In flu and COVID infected mice, nebulized sodium pyruvate decreased morbidity, weight loss, inflammatory cytokines and decreased viral titers compared to placebo controls. The study to be done at Missouri State University is titled ( Two week sub-chronic double-blinded placebo controlled trial designed to determine if sodium pyruvate nasal spray will reduce the symptoms, duration and replication of COVID-19 infection)

DETAILED DESCRIPTION:
Inhibition of Viral Replication, Reduction of the "Cytokine Storm" and reduction of COVID-19 symptoms- Potential Treatment and Preventative for COVID-19

In numerous human clinical trials (17, phase I, II, III clinical trials) submitted to the FDA, with Pulmonary Fibrosis, COPD and Cystic Fibrosis patients, inhaled sodium pyruvate reduced nasal and lung inflammation and congestion by reducing inflammatory cytokines including the IL-6 cytokine that causes the so-called cytokine storm with no known adverse reactions. Cellular Sciences received Orphan Drug Designations for Pulmonary Fibrosis and Cystic Fibrosis. Mice studies conducted by Dr. Lupfer at Missouri State University substantiated our finding by testing nebulized sodium pyruvate in flu (influenza A H1N1 virus) infected mice that decreased morbidity, weight loss, proinflammatory cytokines, and decreased viral titers (virus numbers) compared to the Placebo Control. Additionally, treated mice consumed more chow during infection indicating improved symptoms (same results reported in a pilot mice COVID-19 study). There were notable improvements in pro-inflammatory cytokine production (IL-1β) and lower virus titers (viral numbers) on days 7 post infection in mice treated with Sodium pyruvate compared to the Placebo Control animals. As pyruvate acts on the host immune response, metabolic pathways and not directly on the virus, our data demonstrate that sodium pyruvate is a promising treatment option that is safe, effective, and unlikely to elicit antiviral resistance. Furthermore, we have preliminary data that suggest it may work similarly during other respiratory virus infections including COVID19/SARS-CoV-2.

In a Phase III Placebo Controlled Clinical Trial with Idiopathic Pulmonary Fibrosis Patients, inhaled sodium pyruvate, a Non-Steroidal Nasal Spray (N115) demonstrated a statistically and clinically significant increase in FEV-1, SaO2, FVC, FEV-1/FVC ratios (from 52% to 86%), and a statistically and clinically significant reduction in coughing, hypoxemia and a reduction in nasal and lung inflammation. Inhaled sodium pyruvate alleviated the symptoms associated with the COVID-19 infections in Patients with COPD and Pulmonary Fibrosis. Nasal Nitric Oxide reduces the rate, duration and severity of viral infections in healthy young children and in healthy adults from the Flu, Rhinovirus and Coronavirus. The literature has reported that Nitric Oxide is elicited and inhibits viral replication in pigs infected with porcine respiratory coronavirus. Additionally Nasal Nitric Oxide levels decreases from normal levels found in healthy adults, in patients with asthma (87%), COPD (73%) CF (44%) and Primary Ciliary Dyskinesia (7%). The rate of infections increases with decreasing levels of nasal nitric oxide. Young children, 6-17 years of age, produce (142%) more nitric oxide than healthy adults, which may explain their resistance to COVID-19. Recently, researchers announced that a high percentage of COVID-19 infected patients that were hospitalized were Diabetics or were Pre-Diabetic. The literature has reported that elevated levels of glucose in patients with diabetes mellitus cause a deficiency in the production of nitric oxide by blunting nitric oxide synthesis, which may explain their susceptibility to COVID-19. Sodium pyruvate increases nitric oxide and is safe for use by Patients with Diabetes. The inhalation of nasal sodium pyruvate increased the synthesis of nasal nitric oxide to normal levels in patients with low levels of nitric oxide to increase all lung functions and decrease the rate of infections.

A clinical survey of 367 patients who took a nasal spray similar to EmphyCorp' s N115 formula, over a two-year period demonstrated a statistically significant decrease in the number, symptoms, and severity of seasonal flu respiratory tract infections. The number of flu or colds was reduced by 70% in Children and approximately 52% in Pregnant Women, Patients with Allergic Rhinitis, Diabetes, and Pulmonary Fibrosis. It has been used successfully by over 2 million patients globally in over 200 hospitals during the past 5 years to treat nasal and lung inflammation, congestion in Patients with COPD, Allergic Rhinitis, Pulmonary Fibrosis, sinusitis, the flu and Cystic Fibrosis, with no adverse events reported. It has been used by Children, Diabetics, and Hypertensives, with efficacy and with no known side effects. It has even been shown to be safe for use by Pregnant Women, for whom steroids are contraindicated as they increase the risk of low birth-weight babies.

Proactive treatments with sodium pyruvate are not toxic and could be of benefit to children that are afflicted by many respiratory viruses and as a potential treatment for COVID long haulers.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a confirmed COVID-19 viral infection, as determined by a qualified laboratory test. A nasal swab or saliva test analyzed by qPCR for COVID19.
2. Individuals who agree to abstain from sexual intercourse, or agree to use condoms or vaginal diaphragms or other devices designed to prevent contraception, during the entire course of the study

Exclusion Criteria

1. Viral infections other than COVID-19.
2. Clinically significant cardiac disease including uncontrolled congestive heart failure and unstable angina
3. Pregnancy
4. Females of child bearing potential age not on adequate contraception or lactating
5. Subjects receiving systemic corticosteroid treatment within one month of Screening Visit
6. Subjects Less than 18 years of age
7. Hospitalization within last 6 months due to acute exacerbation of airway disease
8. Subjects with a clinically significant abnormal chest x-ray within past 12 months
9. Medication changes within one month of study entry
10. Subjects who have participated in another investigation drug treatment study within the previous month.
11. Subjects with a current history of alcohol or recreational drug abuse.
12. Subjects who have taken dietary supplements containing pyruvate within 24 hours prior to the screening visit.

Inclusion of Women and Minorities Every attempt will be made to include all genders, and minorities that present with an active COVID-19 infection that are not exempted due to exclusion criteria.

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Amen, Ph.D., Study Director — VP of Regulatory affairs
Locations (2):
- United States (2):
  - Family First Medical Research Center, Virginia Gardens, Florida
  - Missouri State University, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reel JM, Lupfer CR. Sodium Pyruvate Ameliorates Influenza A Virus Infection In Vivo. Microbiology Research. 2021; 12: 258-267.
- [Background] Abusalamah H, Reel JM, Lupfer CR. Pyruvate affects inflammatory responses of macrophages during influenza A virus infection. Virus Res. 2020 Sep;286:198088. doi: 10.1016/j.virusres.2020.198088. Epub 2020 Jul 4. PMID 32634445
- See also: Summary of previous clinical trials for sodium pyruvate — http://emphycorp.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray: In this arm, patients will be provided with N115 sodium pyruvate nasal spray and instructed to use it 3x daily for 14 days. This group will be compared to the placebo control group to determine if sodium pyruvate reduces the symptoms, duration and replication of COVID-19 infections.
  Sodium Pyruvate: Subjects will use a sodium pyruvate nasal spray 3x daily for 14 days.
- Placebo Control Treatment of COVID-19 Infected Patients: In this arm, patients will be provided with a saline nasal spray as a placebo control. Patients will use the saline nasal spray 3x daily for 14 days, similar to the sodium pyruvate drug arm. This will serve as a control for the symptoms, duration and replication of COVID-19 infections.
  Saline: Subjects will use a saline nasal spray 3x daily for 14 days.
Period: Overall Study
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (17.57) | 54.73 (19.51) | 53.97 (18.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Change COVID-19 Viral Titers.
Description: RT-PCR was used to assess viral titers from nasal swabs from COVID19 patients. Swabs were collected and tested every 2 days for 14 days.
Time Frame: Day 0, 2, 4, 6, 8, 10, 12, and 14
Measure: Mean (Standard Error); unit: Log10 viral RNA copies
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 15 | 15
Log10 viral RNA copies
  Day 0 | 5.61 (0.26) | 6.57 (0.24)
  Day 2 | 4.67 (0.26) | 5.86 (0.20)
  Day 4 | 4.27 (0.26) | 5.18 (0.21)
  Day 6 | 3.88 (0.31) | 4.55 (0.22)
  Day 8 | 3.48 (0.34) | 4.11 (0.20)
  Day 10 | 3.18 (0.24) | 3.71 (0.25)
  Day 12 | 2.96 (0.23) | 3.35 (0.34)
  Day 14 | 2.34 (0.11) | 2.78 (0.39)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.0197, ANOVA; two-way ANOVA; Mean Difference (Final Values) = -0.3379, 95% CI 2-sided [-0.6213 to -0.0545], Standard Error of Mean 0.1438

2. Primary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect SaO2 in COVID-19 Infected Patients.
Description: Percent SaO2 was measured every other day by clinic staff.
Time Frame: Day 0, 2, 4, 6, 8, 10, 12, and 14
Measure: Mean (Standard Deviation); unit: % Blood oxygen saturation
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 15 | 15
% Blood oxygen saturation
  Day 0 | 95.73 (0.96) | 95.4 (0.83)
  Day 2 | 95.6 (0.99) | 95.73 (0.59)
  Day 4 | 95.67 (0.82) | 95.8 (0.77)
  Day 6 | 96.07 (1.22) | 96.43 (0.76)
  Day 8 | 96.93 (1.03) | 96.71 (0.91)
  Day 10 | 97.33 (0.82) | 97.21 (0.97)
  Day 12 | 97.53 (0.83) | 97.5 (0.76)
  Day 14 | 97.8 (0.56) | 97.57 (0.76)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.736, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 0.0381, 95% CI 2-sided [-0.1843 to 0.2605], Standard Error of Mean 0.1129

3. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Fever in COVID-19 Infected Patients.
Description: To evaluate the ability of the N115 nasal spray to improve fever in COVID19 patients oral measurement of body temperature was assessed every morning and every evening for 14 days. Reported values are the average daily body temperature.
Time Frame: Twice daily (morning and evening) from Day 1-14
Measure: Mean (Standard Error); unit: Degrees Fahrenheit
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 15 | 15
Degrees Fahrenheit
  Day 1 | 99.72 (0.35) | 99.82 (0.20)
  Day 2 | 100.47 (0.43) | 100.18 (0.42)
  Day 3 | 100.12 (0.22) | 99.51 (0.28)
  Day 4 | 100.09 (0.42) | 99.8 (0.37)
  Day 5 | 100.05 (0.36) | 99.43 (0.30)
  Day 6 | 99.8 (0.33) | 99.37 (0.22)
  Day 7 | 99.47 (0.29) | 98.97 (0.15)
  Day 8 | 99.56 (0.37) | 99.3 (0.15)
  Day 9 | 99.39 (0.28) | 99.17 (0.14)
  Day 10 | 99.4 (0.25) | 99.21 (0.39)
  Day 11 | 99.53 (0.28) | 99.22 (0.20)
  Day 12 | 99.24 (0.16) | 99.05 (0.13)
  Day 13 | 99.17 (0.12) | 98.84 (0.16)
  Day 14 | 99.18 (0.15) | 98.91 (0.13)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.0030, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 0.3131, 95% CI 2-sided [0.1069 to 0.5193], Standard Error of Mean 0.1049

4. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Body Aches in COVID-19 Infected Patients.
Description: Patients self reported the symptom in a patient log daily for 14 days. A Likert scale from 0-10 was used to rank the symptom severity, with 10 representing the most severe symptoms.
Time Frame: Daily from Day 1-14
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 10 | 8
units on a scale
  Day 1 | 6.4 (2.67) | 5.13 (2.85)
  Day 2 | 6.4 (2.67) | 5.13 (2.85)
  Day 3 | 6.4 (2.67) | 4.88 (2.8)
  Day 4 | 6.0 (1.94) | 4.75 (2.6)
  Day 5 | 5.9 (1.79) | 4.25 (2.49)
  Day 6 | 5.5 (2.12) | 4 (2.56)
  Day 7 | 5.3 (2.21) | 3.5 (2.45)
  Day 8 | 5.6 (2.59) | 3.25 (2.6)
  Day 9 | 5 (2.4) | 3.125 (2.42)
  Day 10 | 5 (2.4) | 3 (2.51)
  Day 11 | 4.4 (2.22) | 2.375 (2.56)
  Day 12 | 4.1 (2.08) | 2 (2.39)
  Day 13 | 3.6 (2.27) | 1.75 (1.98)
  Day 14 | 3 (1.83) | 1.63 (1.92)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p < 0.0001, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 1.704, 95% CI 2-sided [1.105 to 2.302], Standard Error of Mean 0.3035

5. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Headaches in COVID-19 Infected Patients.
Description: as for outcome 4
Time Frame: Daily form day 1-14.
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 4 | 7
units on a scale
  Day 1 | 4.25 (3.1) | 3.14 (2.79)
  Day 2 | 4.25 (2.75) | 3.14 (2.79)
  Day 3 | 4.75 (2.22) | 2.86 (2.27)
  Day 4 | 4.25 (2.36) | 2.71 (2.36)
  Day 5 | 4.25 (2.22) | 2.29 (1.89)
  Day 6 | 3.75 (1.89) | 2.14 (2.04)
  Day 7 | 3.75 (2.50) | 2.00 (1.83)
  Day 8 | 3.75 (2.50) | 1.86 (1.95)
  Day 9 | 3.50 (2.38) | 1.57 (1.51)
  Day 10 | 3.00 (1.63) | 1.29 (1.25)
  Day 11 | 3.00 (1.36) | 1.14 (1.07)
  Day 12 | 2.75 (2.22) | 1.00 (1.00)
  Day 13 | 2.75 (1.71) | 1.00 (1.00)
  Day 14 | 2.0 (1.83) | 1.00 (1.00)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p < 0.0001, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 1.633, 95% CI 2-sided [0.9672 to 2.298], Standard Error of Mean 0.3362

6. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Chills in COVID-19 Infected Patients.
Description: as for outcome 4
Time Frame: Daily from day 1-14.
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 8 | 8
units on a scale
  Day 1 | 5 (2.67) | 3.75 (1.67)
  Day 2 | 5.25 (2.55) | 3.50 (2.07)
  Day 3 | 5.25 (2.05) | 3.50 (2.07)
  Day 4 | 4.38 (2.33) | 3.13 (1.96)
  Day 5 | 4.50 (2.33) | 2.75 (1.91)
  Day 6 | 4.00 (2.00) | 2.63 (1.69)
  Day 7 | 4.13 (2.17) | 2.25 (1.28)
  Day 8 | 4.25 (2.12) | 1.75 (1.49)
  Day 9 | 3.88 (2.03) | 1.38 (1.30)
  Day 10 | 3.63 (1.92) | 1.00 (1.07)
  Day 11 | 3.13 (1.81) | 0.75 (1.04)
  Day 12 | 2.88 (1.89) | 0.38 (0.52)
  Day 13 | 2.38 (2.13) | 0.38 (0.52)
  Day 14 | 2.38 (2.13) | 0.38 (0.52)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p < 0.0001, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 1.964, 95% CI 2-sided [1.477 to 2.452], Standard Error of Mean 0.2473

7. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Coughing and Sneezing in COVID-19 Infected Patients.
Description: Patients self reported the symptom in a patient log daily for 14 days. A Likert scale from 0-10 was used to rank the symptom severity, with 10 representing the most severe symptoms. The symptoms of both coughing and sneezing were assessed on the same Likert scale for this Outcome Measure.
Time Frame: Daily from day 1-14.
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 10 | 11
units on a scale
  Day 1 | 3.90 (2.69) | 4.45 (2.16)
  Day 2 | 3.70 (2.58) | 4.45 (2.16)
  Day 3 | 3.50 (2.42) | 4.18 (2.44)
  Day 4 | 3.40 (1.78) | 4.18 (2.27)
  Day 5 | 3.20 (1.93) | 3.64 (2.16)
  Day 6 | 3.10 (2.02) | 3.64 (2.25)
  Day 7 | 2.80 (1.93) | 3.55 (2.16)
  Day 8 | 2.70 (2.0) | 2.82 (2.40)
  Day 9 | 2.40 (1.96) | 2.73 (2.10)
  Day 10 | 190 (1.52) | 2.36 (2.16)
  Day 11 | 1.40 (1.65) | 2.09 (2.17)
  Day 12 | 1.40 (1.65) | 1.64 (1.69)
  Day 13 | 1.10 (1.66) | 1.45 (1.44)
  Day 14 | 1.10 (1.66) | 1.18 (1.17)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.0435, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = -0.4831, 95% CI 2-sided [-0.9521 to -0.01413], Standard Error of Mean 0.2382

8. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Sore Throat in COVID-19 Infected Patients.
Description: as for outcome 4
Time Frame: Daily from day 1-14.
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 7 | 7
units on a scale
  Day 1 | 4.71 (2.29) | 4.71 (1.70)
  Day 2 | 4.71 (2.14) | 4.71 (1.70)
  Day 3 | 4.57 (1.81) | 4.57 (1.72)
  Day 4 | 4.29 (2.06) | 4.57 (1.51)
  Day 5 | 4.14 (2.04) | 4.0 (1.73)
  Day 6 | 4.29 (2.06) | 3.86 (1.77)
  Day 7 | 4.14 (2.12) | 3.71 (1.60)
  Day 8 | 3.29 (2.43) | 3.00 (2.31)
  Day 9 | 2.86 (2.12) | 2.86 (2.12)
  Day 10 | 2.29 (1.70) | 2.57 (2.07)
  Day 11 | 2.00 (1.91) | 2.14 (2.27)
  Day 12 | 1.57 (1.72) | 1.71 (1.60)
  Day 13 | 0.86 (1.46) | 1.57 (1.51)
  Day 14 | 0.86 (1.46) | 1.29 (1.60)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.8509, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = -0.05102, 95% CI 2-sided [-0.5862 to 0.4841], Standard Error of Mean 0.2711

9. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Congestions in COVID-19 Infected Patients.
Description: as for outcome 4
Time Frame: Daily from day 1-14.
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 8 | 10
units on a scale
  Day 1 | 5.00 (3.38) | 5.00 (3.56)
  Day 2 | 5.00 (2.83) | 5.00 (3.62)
  Day 3 | 4.75 (2.92) | 4.90 (3.63)
  Day 4 | 4.50 (2.39) | 4.60 (2.91)
  Day 5 | 3.50 (2.00) | 4.10 (2.85)
  Day 6 | 3.50 (2.00) | 4.30 (2.98)
  Day 7 | 3.25 (1.98) | 3.70 (2.67)
  Day 8 | 4.31 (2.30) | 2.80 (2.74)
  Day 9 | 3.00 (2.39) | 2.60 (2.50)
  Day 10 | 2.88 (1.73) | 2.20 (2.74)
  Day 11 | 2.13 (1.96) | 1.60 (2.07)
  Day 12 | 1.50 (1.31) | 1.50 (2.01)
  Day 13 | 1.00 (1.07) | 0.60 (1.07)
  Day 14 | 1.25 (1.28) | 0.60 (1.07)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.6738, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 0.1339, 95% CI 2-sided [-0.4921 to 0.7600], Standard Error of Mean 0.3177

10. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Trouble Breathing in COVID-19 Infected Patients.
Description: as for outcome 4
Time Frame: Daily from day 1-14
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 12 | 11
units on a scale
  Day 1 | 5.08 (3.73) | 5.18 (4.00)
  Day 2 | 5.25 (3.57) | 5.18 (4.00)
  Day 3 | 5.00 (3.28) | 4.91 (4.04)
  Day 4 | 4.42 (2.71) | 4.27 (3.47)
  Day 5 | 4.17 (2.55) | 4.00 (3.22)
  Day 6 | 3.75 (2.49) | 4.18 (2.99)
  Day 7 | 3.67 (2.35) | 3.55 (2.42)
  Day 8 | 3.67 (2.35) | 3.00 (1.90)
  Day 9 | 2.92 (2.31) | 2.55 (1.75)
  Day 10 | 2.58 (1.51) | 2.00 (1.73)
  Day 11 | 2.17 (1.27) | 1.64 (1.21)
  Day 12 | 1.50 (1.24) | 0.91 (0.83)
  Day 13 | 1.25 (1.06) | 0.36 (0.50)
  Day 14 | 0.92 (1.16) | 0.27 (0.47)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p = 0.2753, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = 0.3095, 95% CI 2-sided [-0.2478 to 0.8669], Standard Error of Mean 0.2832

11. Secondary Outcome: Evaluate the Ability of Inhaled Nasal Sodium Pyruvate to Affect Fatigue in COVID-19 Infected Patients.
Description: as for outcome 4
Time Frame: Daily from day 1-14.
Population: Only patients that reported experiencing this symptom were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
Number analyzed (Participants) | 7 | 4
units on a scale
  Day 1 | 6.43 (1.51) | 7.50 (1.29)
  Day 2 | 6.43 (1.51) | 7.50 (1.29)
  Day 3 | 6.00 (1.91) | 7.25 (1.50)
  Day 4 | 4.86 (1.35) | 7.00 (1.41)
  Day 5 | 4.57 (1.72) | 7.00 (1.41)
  Day 6 | 4.71 (1.50) | 6.50 (2.08)
  Day 7 | 4.57 (1.72) | 6.50 (1.73)
  Day 8 | 4.29 (1.98) | 6.50 (1.73)
  Day 9 | 3.43 (1.90) | 4.50 (1.29)
  Day 10 | 3.29 (1.60) | 4.25 (1.50)
  Day 11 | 2.57 (1.51) | 3.50 (1.91)
  Day 12 | 2.00 (1.00) | 3.50 (1.91)
  Day 13 | 1.57 (1.27) | 2.50 (1.29)
  Day 14 | 1.57 (1.27) | 2.25 (1.26)
Statistical Analysis 1: Comparison: Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray vs Placebo Control Treatment of COVID-19 Infected Patients; Test type: Superiority; p < 0.0001, ANOVA; Two-way ANOVA; Mean Difference (Final Values) = -1.426, 95% CI 2-sided [-1.948 to -0.9043], Standard Error of Mean 0.2636

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Treatment of COVID-19 Infected Patients With a Sodium Pyruvate Nasal Spray | Placebo Control Treatment of COVID-19 Infected Patients
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The number of patients enrolled in this trial was small, thus decreasing the power of the statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT04824365/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04824365/ICF_000.pdf